CLINICAL TRIAL: NCT03717350
Title: A suPAR Guided Double-blind Randomized Clinical Trial of Initiation of Antibiotics for Presumed Infection at the Emergency Department
Brief Title: suPAR to Guide Antibiotics in Emergency Department
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUPERIOR
Record Dates: First submitted 2018-10-20; First posted 2018-10-24 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Sepsis
Keywords: biomarkers; suPAR; outcome; antibiotics
MeSH Terms: conditions — Sepsis | interventions — Meropenem; Carbapenems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Similar appearance of study drug of both arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 100ml of sodium chloride 0.9% within 15 minutes intravenously
  Interventions: Drug: Placebo
- Antibiotic (Active Comparator): 2g of meropenem diluted in 100ml of sodium chloride 0.9% within 15 minutes intravenously
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — 2g of meropenem diluted in 100ml of sodium chloride 0.9% within 15 minutes intravenously administered once
  Other Names: Carbapenem
  Arms: Antibiotic
Drug: Placebo — 100ml of sodium chloride 0.9% within 15 minutes intravenously once
  Other Names: Diluent
  Arms: Placebo

SUMMARY:
The aim of the current study is to evaluate suPAR - guided medical intervention, consisting of early antibiotic administration at the emergency room for presumed infection and sepsis and evaluate the impact of this intervention to the patients' final outcome. Since the traditionally used biomarkers (PCT, CRP) and scores (SOFA score) for early recognition of severity of infection fail to achieve maximum accuracy in all cases, suPAR levels are assessed as a probably better prognostic rule for early recognition of severe infections. The primary study endpoint will be the comparative efficacy of the early suPAR-guided administration of antibiotics versus standard practice on 28-day mortality.

DETAILED DESCRIPTION:
Sepsis is among the leading causes of death worldwide. It is well-perceived that early recognition of sepsis is the mainstay of treatment. Recently it has been proposed that the quick sequential organ fialure assessment (qSOFA) score can be used as a screening tool in the emergency department (ED) to triage patients with high-risk of death; patients scoring positive at least two of the three signs of qSOFA are at a high-risk for death. However, this is challenged since it may be the case that the risk of death is high even among patients with only one sign of qSOFA.

Soluble urokinase plasminogen activator receptor (suPAR), the soluble form of the membrane bound receptor (uPAR), is a recently known glycoprotein involved in inflammation. uPAR is expressed on various immune cells (neutrophils, lymphocytes, monocytes, macrophages) and is cleaved from their surface after an inflammatory stimuli to enhance chemotaxis and cell migration. Increased suPAR blood levels mirror the degree of activation of the immune system by different antigenic stimuli including diverse neoplastic and infectious agents and other inflammation-mediated diseases. SuPAR levels generally correlate to the severity of the disease.

It has been shown that suPAR blood levels have low diagnostic value (cannot discriminate between bacterial, viral or parasitic infection, Gram (+) or Gram (-) bacteraemia. However, they present superior prognostic value as compared with single parameters of inflammation and organ dysfunction (like C-reactive protein (CRP) and procalcitonin (PCT) in critically ill patients, and suPAR's prognostic value of death is even more enhanced when combined to other biomarkers and physiological scores (e.g. Acute Physiology and Chronic Health Evaluation-APACHE II).

Why choose suPAR as biomarker at emergency basis? Because, in contrast to many pro-inflammatory cytokines, suPAR exhibits favorable properties due to its high stability in serum samples and limited circadian changes in plasma concentrations. It also constitutes a serum/plasma biomarker that is easily performed on-site and provides information within one hour after sampling21, 22.

Unpublished data of the Hellenic Sepsis Study Group (HSSG) suggest that among patients with at least one sign of the qSOFA score, those with suPAR greater than 12 ng/ml are at a substantial risk for death with mortality exceeding 30%. To this end, patients with suspicion for an infection and with qSOFA 1 and suPAR greater than 12 ng/ml constitute a group of patients requiring early intervention.

The aim of the current study is to evaluate suPAR - guided medical intervention, consisting of early antibiotics' administration at the emergency room for presumed infection and sepsis and evaluate the impact of this intervention to the patients' final outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by the patient or by their legal representative in case of patients unable to consent
2. Age equal to or above 18 years
3. Male or female gender
4. Clinical suspicion of infection
5. qSOFA equal to 1 point
6. suPAR blood level equal or above 12 ng/ml

Exclusion Criteria:

1. Denial to consent
2. Patients with 2 or 3 qSOFA signs
3. Pregnancy (confirmed by blood or urinary pregnancy test) for female patients of reproductive age
4. Organ transplantation
5. Fully-blown sepsis with overt failing organs necessitating immediate resuscitation as defined by the attending physicians
6. Do not resuscitate decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-10-27 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the applied intervention versus standard practice on the early worsening of the patient. | 1 day (24 hours)
  The primary study endpoint will be the comparative efficacy of the applied intervention (meropenem versus standard practice on the early worsening of the patient. This is defined as any at least one point increase of the admission total SOFA score the first 24 hours.

SECONDARY OUTCOMES:
Sepsis mortality | 28 days
  Comparative efficacy of the applied intervention on mortality for patients meeting the Sepsis-3 definition of sepsis
Short-term mortality | 7 days
  Comparative efficacy of the applied intervention on 7-day mortality
Long-term mortality 1 | 60 days
  Comparative efficacy of the applied intervention on 60-day mortality
Long-term mortality 2 | 90 days
  Comparative efficacy of the applied intervention on 90-day mortality
Infection resolution | 90 days
  Effect of the intervention on the time to infection resolution. This time point is limited for patients who will eventually be diagnosed of a specific infectious diseases making them eligible for the study and it is defined as the time point when all clinical signs of the infection are cleared.
Change of initial treatment | 28 days
  Comparative efficacy of the applied intervention on the need to change antibiotics
Duration of hospitalization | 90 days
  Comparative efficacy of the applied intervention on the duration of hospitalization
Rate of new infections | 90 days
  Comparative efficacy of the applied intervention on the rate of new infections
The early worsening of the patient | 1 day (24 hours)
  The early worsening of the patient defined as for the primary endpoint but analyzed separately per quartile of the total SOFA score of the patient population

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — Attikon Hospital
Locations (5):
- Greece (5):
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens, Attica
  - 1st Department of Internal Medicine of G. GENNIMATAS General Hospital, Athens
  - 3rd Department of Internal Medicine at SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - Εmergency Department of Sismanogleion Athens General Hospital, Athens
  - Department of Internal Medicine, Patras University Hospital, Pátrai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ, Tsaganos T, Tsangaris I, Lada M, Routsi C, Sinapidis D, Koupetori M, Bristianou M, Adamis G, Mandragos K, Dalekos GN, Kritselis I, Giannikopoulos G, Koutelidakis I, Pavlaki M, Antoniadou E, Vlachogiannis G, Koulouras V, Prekates A, Dimopoulos G, Koutsoukou A, Pnevmatikos I, Ioakeimidou A, Kotanidou A, Orfanos SE, Armaganidis A, Gogos C; Hellenic Sepsis Study Group. Validation of the new Sepsis-3 definitions: proposal for improvement in early risk identification. Clin Microbiol Infect. 2017 Feb;23(2):104-109. doi: 10.1016/j.cmi.2016.11.003. Epub 2016 Nov 14. PMID 27856268
- [Background] Giamarellos-Bourboulis EJ, Norrby-Teglund A, Mylona V, Savva A, Tsangaris I, Dimopoulou I, Mouktaroudi M, Raftogiannis M, Georgitsi M, Linner A, Adamis G, Antonopoulou A, Apostolidou E, Chrisofos M, Katsenos C, Koutelidakis I, Kotzampassi K, Koratzanis G, Koupetori M, Kritselis I, Lymberopoulou K, Mandragos K, Marioli A, Sunden-Cullberg J, Mega A, Prekates A, Routsi C, Gogos C, Treutiger CJ, Armaganidis A, Dimopoulos G. Risk assessment in sepsis: a new prognostication rule by APACHE II score and serum soluble urokinase plasminogen activator receptor. Crit Care. 2012 Aug 8;16(4):R149. doi: 10.1186/cc11463. PMID 22873681
- [Derived] Adami ME, Kotsaki A, Antonakos N, Giannitsioti E, Chalvatzis S, Saridaki M, Avgoustou C, Akinosoglou K, Dakou K, Damoraki G, Katrini K, Koufargyris P, Lekakis V, Panagaki A, Safarika A, Eugen-Olsen J, Giamarellos-Bourboulis EJ. qSOFA combined with suPAR for early risk detection and guidance of antibiotic treatment in the emergency department: a randomized controlled trial. Crit Care. 2024 Feb 6;28(1):42. doi: 10.1186/s13054-024-04825-2. PMID 38321472
- [Derived] Kyriazopoulou E, Poulakou G, Giamarellos-Bourboulis EJ. Biomarkers in sepsis: can they help improve patient outcome? Curr Opin Infect Dis. 2021 Apr 1;34(2):126-134. doi: 10.1097/QCO.0000000000000707. PMID 33534419